CLINICAL TRIAL: NCT00168844
Title: A Randomised, Double-Blind, Placebo-Controlled, Parallel-Group Efficacy and Safety Comparison of One-Year Treatment of Two Doses (5mg and 10mg) of Tiotropium Inhalation Solution Delivered by the Respimat Device in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Tiotropium / Respimat One-Year Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 205.254
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Results first posted 2009-10-07 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2013-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

ARMS (3):
- Tiotropium Respimat 5mcg (Tio R5) (Other)
  Interventions: Drug: Tiotropium Inhalation Solution
- Tiotropium Respimat 10mcg (Tio R10) (Other)
  Interventions: Drug: Tiotropium Inhalation Solution
- Placebo (Other)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Tiotropium Inhalation Solution
  Arms: Tiotropium Respimat 10mcg (Tio R10); Tiotropium Respimat 5mcg (Tio R5)
Other: Placebo
  Arms: Placebo

SUMMARY:
To evaluate the long term effects of treatment with two doses of Tiotropium delivered by the Respimat inhaler in patients with COPD.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 983 (Actual)
Dates: Start 2003-01; Primary Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (72):
- United States (12):
  - Boehringer Ingelheim Investigational Site, Los Angeles, California
  - Boehringer Ingelheim Investigational Site, Pismo Beach, California
  - Boehringer Ingelheim Investigational Site, San Diego, California
  - Boehringer Ingelheim Investigational Site, Fort Collins, Colorado
  - Boehringer Ingelheim Investigational Site, Minneapolis, Minnesota
  - Boehringer Ingelheim Investigational Site, Larchmont, New York
  - Boehringer Ingelheim Investigational Site, Raleigh, North Carolina
  - Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - Boehringer Ingelheim Investigational Site, Harker Heights, Texas
  - Boehringer Ingelheim Investigational Site, Houston, Texas
  - Boehringer Ingelheim Investigational Site, Fredericksburg, Virginia
  - Boehringer Ingelheim Investigational Site, Harrisonburg, Virginia
- Australia (5):
  - Boehringer Ingelheim Investigational Site, Toorak Gardens, South Australia
  - Boehringer Ingelheim Investigational Site, Woodville, South Australia
  - Boehringer Ingelheim Investigational Site, Clayton, Victoria
  - Boehringer Ingelheim Investigational Site, Frankston, Victoria
  - Boehringer Ingelheim Investigational Site, Perth, Western Australia
- Belgium (6):
  - Boehringer Ingelheim Investigational Site, Antwerp
  - Boehringer Ingelheim Investigational Site, Brussels
  - Boehringer Ingelheim Investigational Site, Genk
  - Boehringer Ingelheim Investigational Site, Ghent
  - Boehringer Ingelheim Investigational Site, Liège
  - Boehringer Ingelheim Investigational Site, Wavre
- Canada (7):
  - Boehringer Ingelheim Investigational Site, Edmonton, Alberta
  - Boehringer Ingelheim Investigational Site, Halifax, Nova Scotia
  - Boehringer Ingelheim Investigational Site, Courtice, Ontario
  - Boehringer Ingelheim Investigational Site, Mississauga, Ontario
  - Boehringer Ingelheim Investigational Site, Ottawa, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - Boehringer Ingelheim Investigational Site, Sainte-Foy, Quebec
- France (5):
  - Boehringer Ingelheim Investigational Site, Angers
  - Boehringer Ingelheim Investigational Site, Beuvry
  - Boehringer Ingelheim Investigational Site, Cambrai
  - Boehringer Ingelheim Investigational Site, Lille
  - Boehringer Ingelheim Investigational Site, Metz
- Germany (5):
  - Boehringer Ingelheim Investigational Site, Berlin
  - Boehringer Ingelheim Investigational Site, Darmstadt
  - Boehringer Ingelheim Investigational Site, Gelnhausen
  - Boehringer Ingelheim Investigational Site, Kassel
  - Boehringer Ingelheim Investigational Site, Rüdersdorf
- Greece (5):
  - Boehringer Ingelheim Investigational Site, Athens
  - Boehringer Ingelheim Investigational Site, Heraklion
  - Boehringer Ingelheim Investigational Site, Larissa
  - Boehringer Ingelheim Investigational Site, Maroussi, Athens
  - Boehringer Ingelheim Investigational Site, Melissia-Athens
- Netherlands (6):
  - Boehringer Ingelheim Investigational Site, Breda
  - Boehringer Ingelheim Investigational Site, Dordrecht
  - Boehringer Ingelheim Investigational Site, Groningen
  - Boehringer Ingelheim Investigational Site, Harderwijk
  - Boehringer Ingelheim Investigational Site, Heerlen
  - Boehringer Ingelheim Investigational Site, Zutphen
- Norway (3):
  - Boehringer Ingelheim Investigational Site, Ålesund
  - Boehringer Ingelheim Investigational Site, Oslo
  - Boehringer Ingelheim Investigational Site, Trondheim
- Boehringer Ingelheim Investigational Site, Moscow, Russia
- Spain (4):
  - Boehringer Ingelheim Investigational Site, Alicante
  - Boehringer Ingelheim Investigational Site, Las Palmas de Gran Canaria
  - Boehringer Ingelheim Investigational Site, Madrid
  - Boehringer Ingelheim Investigational Site, Vic (Barcelona)
- Sweden (4):
  - Boehringer Ingelheim Investigational Site, Motala
  - Boehringer Ingelheim Investigational Site, Skövde
  - Boehringer Ingelheim Investigational Site, Uppsala
  - Boehringer Ingelheim Investigational Site, Varberg
- Turkey (Türkiye) (3):
  - Boehringer Ingelheim Investigational Site, Ankara
  - Boehringer Ingelheim Investigational Site, Bursa
  - Boehringer Ingelheim Investigational Site, Istanbul
- United Kingdom (6):
  - Boehringer Ingelheim Investigational Site, Birmingham
  - Boehringer Ingelheim Investigational Site, Bristol
  - Boehringer Ingelheim Investigational Site, Nottingham
  - Boehringer Ingelheim Investigational Site, Sheffield
  - Boehringer Ingelheim Investigational Site, Swansea
  - Boehringer Ingelheim Investigational Site, Torquay

REFERENCES:
- [Derived] Singh D, Wedzicha JA, Siddiqui S, de la Hoz A, Xue W, Magnussen H, Miravitlles M, Chalmers JD, Calverley PMA. Blood eosinophils as a biomarker of future COPD exacerbation risk: pooled data from 11 clinical trials. Respir Res. 2020 Sep 17;21(1):240. doi: 10.1186/s12931-020-01482-1. PMID 32943047
- [Derived] Hohlfeld JM, Furtwaengler A, Konen-Bergmann M, Wallenstein G, Walter B, Bateman ED. Cardiac safety of tiotropium in patients with COPD: a combined analysis of Holter-ECG data from four randomised clinical trials. Int J Clin Pract. 2015 Jan;69(1):72-80. doi: 10.1111/ijcp.12596. Epub 2014 Dec 11. PMID 25496316
- [Derived] Hodder R, Pavia D, Lee A, Bateman E. Lack of paradoxical bronchoconstriction after administration of tiotropium via Respimat(R) Soft Mist Inhaler in COPD. Int J Chron Obstruct Pulmon Dis. 2011;6:245-51. doi: 10.2147/COPD.S16094. Epub 2011 Apr 26. PMID 21814460

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Feb 2003 - Jun 2004, hospital and primary care clinics
Groups:
- Tiotropium Respimat 5mcg (Tio R5): Tiotropium Bromide inhalation solution delivered from Respimat Inhaler (5 mcg)
- Tiotropium Respimat 10mcg (Tio R10): Tiotropium Bromide inhalation solution delivered from Respimat Inhaler (10 mcg)
- Placebo: Placebo inhalation solution delivered from Respimat Inhaler (matching placebo)
Period: Overall Study
Arm/Group | Tiotropium Respimat 5mcg (Tio R5) | Tiotropium Respimat 10mcg (Tio R10) | Placebo
Started | 332 | 332 | 319
Completed | 277 | 277 | 228
Not Completed | 55 | 55 | 91
Not completed — Adverse Event | 31 | 32 | 48
Not completed — Lost to Follow-up | 4 | 5 | 11
Not completed — Withdrawal by Subject | 12 | 9 | 19
Not completed — Protocol Violation | 2 | 2 | 4
Not completed — Other | 6 | 7 | 9

BASELINE CHARACTERISTICS:
Groups:
- Tiotropium Respimat 5mcg: Tiotropium Bromide inhalation solution delivered from Respimat Inhaler (5 mcg)
- Tiotropium Respimat 10mcg: Tiotropium Bromide inhalation solution delivered from Respimat Inhaler (10 mcg)
- Total: Total of all reporting groups
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo | Total
Number analyzed (Participants) | 332 | 332 | 319 | 983
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (8.2) | 64.6 (8.4) | 64.7 (8.9) | 64.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 80 | 67 | 236
  Male | 243 | 252 | 252 | 747

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 at Week 48, Full Analysis Set - Clinic Spirometry (FAS-PFT)
Description: Trough Forced Expiratory Volume in 1 second (FEV1)
Time Frame: 10 minutes prior to test-drug inhalation and at 5, 30 and 60 minutes and 2 and 3 hours after inhalation of study medication
Population: Full Analysis Set - Clinic Spirometry (FAS-PFT)
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 326 | 320 | 296
Litres | 0.097 (0.013) | 0.116 (0.014) | -0.046 (0.014)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry,centre and baseline value; Mean Difference (Final Values) = 0.142, Standard Error of Mean 0.019 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry,centre and baseline value; Mean Difference (Final Values) = 0.161, Standard Error of Mean 0.020 — Tiotropium Respimat 10mcg - Placebo

2. Primary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Total Score, Full Analysis Set - Saint George's Respiratory Questionnaire (FAS-QOL)
Description: Rating scale of 3 domains - symptoms, activities and impact (weighted). Worst score = 100, best score = 0
Time Frame: Week 48
Population: Full Analysis Set - Saint George's Respiratory Questionnaire (FAS-QOL)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 318 | 315 | 275
Points on a scale | 39.648 (0.676) | 38.675 (0.679) | 42.917 (0.728)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Test type: Superiority or Other; p = 0.0011, ANCOVA; The means are adjusted for centre, smoking status at entry and baseline value; Mean Difference (Final Values) = -3.269, Standard Error of Mean 0.996 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The means are adjusted for centre, smoking status at entry and baseline value; Mean Difference (Final Values) = -4.242, Standard Error of Mean 0.999 — Tiotropium Respimat 10mcg - Placebo

3. Primary Outcome: TDI Focal Score, Full Analysis Set - Transitional Dyspnoea Index (FAS-TDI) (Combined Studies)
Description: Rating scale of 3 components - change in functional impairment, change in magnitude of tasks, change in magnitude of efforts. Worst score = -9, best score = +9
  For this endpoint data of twin studies NCT00168844 and NCT00168831 was combined.
Time Frame: Week 48
Population: Full Analysis Set - Transitional Dyspnoea Index (FAS-TDI)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 628 | 618 | 552
Points on a scale | 1.890 (0.112) | 1.913 (0.113) | 0.837 (0.120)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The means are adjusted for centre, smoking status at entry and baseline value; Mean Difference (Final Values) = 1.053, Standard Error of Mean 0.165 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA; The means are adjusted for centre, smoking status at entry and baseline value; Mean Difference (Final Values) = 1.075, Standard Error of Mean 0.166

4. Primary Outcome: COPD Exacerbation Rate, Safety Set (SS) (Combined Studies)
Description: Number of Chronic Obstructive Pulmonary Disease (COPD) exacerbations per patient year.
  For this endpoint data of the twin studies NCT00168844 and NCT00168831 was combined.
Time Frame: 48 weeks
Population: Safety Set. Combined analysis of studies NCT00168844 and NCT00168831. 670 patients analysed in total comprises 338 patients from NCT00168831 and 332 patients from study NCT00168844, 667 patients - 335 and 332, 653 patients - 334 and 319 respectively.
Measure: Mean (Standard Deviation); unit: Number of exacerbations per patient year
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 670 | 667 | 653
Number of exacerbations per patient year | 0.93 (2.02) | 1.02 (3.05) | 1.91 (8.17)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Test type: Superiority or Other; p = 0.0002, Poisson regression; Odds Ratio (OR) = 0.782, 95% CI 2-sided [0.687 to 0.890] — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Test type: Superiority or Other; p < 0.0001, Poisson regression; Odds Ratio (OR) = 0.725, 95% CI 2-sided [0.635 to 0.828] — Tiotropium Respimat 10mcg - Placebo

5. Secondary Outcome: Change From Baseline in Heart Rate
Description: Week 40 pre-dose - baseline
Time Frame: Baseline to Week 40 pre-dose
Population: Combined analysis of studies NCT00168844 and NCT00168831 in subset of patients who had additional 12-lead electrocardiogram (ECG) and 24-hour Holter monitoring performed (see protocol and clinical trial report)
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 155 | 135 | 109
beats per minute (bpm) | 2.1 (12.4) | 3.6 (10.5) | 1.8 (9.7)

6. Secondary Outcome: Change From Baseline in PR Interval
Time Frame: Baseline to Week 40 pre-dose
Population: Combined analysis of studies NCT00168844 and NCT00168831 in subset of patients who had additional 12-lead ECG and 24-hour Holter monitoring performed (see protocol and clinical trial report)
Measure: Mean (Standard Deviation); unit: milliseconds (msec)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 150 | 131 | 105
milliseconds (msec) | -0.8 (20.2) | -2.5 (15.1) | -0.5 (15.3)

7. Secondary Outcome: Change From Baseline in QRS Interval
Description: Week 40 pre-dose - baseline
Time Frame: Baseline to Week 40 pre-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 155 | 135 | 109
msec | 0.9 (9.4) | 1.7 (12.1) | -1.1 (10.3)

8. Secondary Outcome: Change From Baseline in QT Interval
Description: Week 40 pre-dose - baseline
Time Frame: Baseline to Week 40 pre-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 155 | 135 | 109
msec | -4.6 (26.5) | -3.5 (25.2) | -3.2 (22.3)

9. Secondary Outcome: Change From Baseline in QT Interval (Bazett)
Description: Week 40 pre-dose - baseline
Time Frame: Baseline to Week 40 pre-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 155 | 135 | 109
msec | -0.5 (29.9) | 5.4 (24.0) | 2.5 (23.4)

10. Secondary Outcome: Change From Baseline in QT Interval (Fridericia)
Description: Week 40 pre-dose - baseline
Time Frame: Baseline to Week 40 pre-dose
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 155 | 135 | 109
msec | -2.0 (24.3) | 2.2 (21.3) | 0.5 (19.5)

11. Secondary Outcome: Change From Baseline in Heart Rate
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
bpm | 0.3 (5.4) | 1.2 (6.4) | 0.3 (6.6)

12. Secondary Outcome: Change From Baseline in Supraventricular Premature Beat (SVPB) Total
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: premature beats per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
premature beats per 24 hours | -3.4 (94.2) | 6.8 (87.4) | 20.9 (125.8)

13. Secondary Outcome: Holter (24-hour Period) - SVPB (Supraventricular Premature Beat) Run Events Change From Baseline in Supraventricular Premature Beat (SVPB) Run Events
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: events per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
events per 24 hours | 0.0 (0.6) | -0.1 (0.5) | -0.1 (1.6)

14. Secondary Outcome: Change From Baseline in SVPB Pairs
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pairs per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
pairs per 24 hours | -0.4 (4.0) | -0.2 (2.3) | 2.0 (16.4)

15. Secondary Outcome: Change From Baseline in Ventricular Premature Beat (VPB) Total
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: premature beats per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
premature beats per 24 hours | -14.3 (105.9) | 4.6 (68.8) | -24.1 (182.3)

16. Secondary Outcome: Change From Baseline in VPB Run Events
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: events per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
events per 24 hours | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.0)

17. Secondary Outcome: Change From Baseline in VPB Pairs
Description: Week 40 - baseline
Time Frame: Baseline to Week 40
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pairs per 24 hours
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 77 | 66 | 56
pairs per 24 hours | -0.2 (1.6) | -0.1 (3.8) | -0.9 (5.7)

18. Secondary Outcome: Change From Baseline in Haematocrit, Packed Cell Volume (PCV)
Description: Volume of red cells (erythrocytes) in blood, expressed as a fraction (percentage) of the total volume of blood
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: Percentage of erythrocytes
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 280 | 282 | 244
Percentage of erythrocytes | 0 (4) | -1 (4) | 0 (4)

19. Secondary Outcome: Change From Baseline in Haemoglobin
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: grams per litre (g/L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 291 | 289 | 255
grams per litre (g/L) | -1 (10) | -2 (11) | 1 (12)

20. Secondary Outcome: Change From Baseline in Red Blood Cell Count
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^12/Litre (L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 291 | 289 | 254
10^12/Litre (L) | 0.0 (0.3) | -0.1 (0.3) | 0.0 (0.3)

21. Secondary Outcome: Change From Baseline in White Blood Cell Count
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/Litre (L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 291 | 289 | 255
10^9/Litre (L) | 0.1 (1.4) | 0.0 (1.5) | 0.2 (1.5)

22. Secondary Outcome: Change From Baseline in Platelets
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 280 | 250
10^9/L | 4 (30) | 1 (31) | 7 (30)

23. Secondary Outcome: Change From Baseline in Neutrophils
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 289 | 254
percentage of white blood cell count | 1 (8) | 1 (8) | 1 (8)

24. Secondary Outcome: Change From Baseline in Eosinophils
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 289 | 254
percentage of white blood cell count | 0 (2) | 0 (2) | 0 (2)

25. Secondary Outcome: Change From Baseline in Basophils
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 289 | 254
percentage of white blood cell count | 0 (0) | 0 (0) | 0 (0)

26. Secondary Outcome: Change From Baseline in Lymphocytes
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 289 | 254
percentage of white blood cell count | -1 (4) | -1 (4) | 0 (4)

27. Secondary Outcome: Change From Baseline in Monocytes
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: percentage of white blood cell count
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 289 | 254
percentage of white blood cell count | 0 (4) | 0 (3) | 0 (4)

28. Secondary Outcome: Change From Baseline in Neutrophils (Absolute)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 289 | 254
10^9/L | 0.2 (1.5) | 0.1 (1.6) | 0.2 (1.6)

29. Secondary Outcome: Change From Baseline in Lymphocytes (Absolute)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 289 | 254
10^9/L | 0.0 (0.6) | -0.1 (0.7) | 0.1 (0.6)

30. Secondary Outcome: Change From Baseline in Eosinophils (Absolute)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 289 | 254
10^9/L | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.1)

31. Secondary Outcome: Change From Baseline in Basophils (Absolute)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 289 | 254
10^9/L | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.0)

32. Secondary Outcome: Change From Baseline in Monocytes (Absolute)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: 10^9/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 288 | 289 | 254
10^9/L | 0.0 (0.2) | 0.0 (0.2) | 0.0 (0.2)

33. Secondary Outcome: Change From Baseline in Calcium
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: millimoles per litre (mmol/L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 289 | 295 | 259
millimoles per litre (mmol/L) | 0.0 (0.1) | 0.0 (0.1) | 0.0 (0.2)

34. Secondary Outcome: Change From Baseline in Phosphate
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 291 | 296 | 261
mmol/L | 0.02 (0.25) | 0.00 (0.23) | 0.01 (0.23)

35. Secondary Outcome: Change From Baseline in Aspartate Transaminase (AST)/Glutamic-Oxaloacetic Transaminase (GOT), Serum GOT (SGOT)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: Units per litre (U/L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 292 | 296 | 261
Units per litre (U/L) | -3 (17) | -1 (13) | 0 (17)

36. Secondary Outcome: Change From Baseline in Alanine Transaminase (ALT)/Glutamic Pyruvic Transaminase (GPT), Serum GPT (SGPT)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 292 | 296 | 261
U/L | -2 (13) | -1 (15) | -1 (15)

37. Secondary Outcome: Change From Baseline in Alkaline Phosphatase
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 290 | 295 | 259
U/L | -3 (21) | -6 (20) | -5 (27)

38. Secondary Outcome: Change From Baseline in Lactic Dehydrogenase (LDH)
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 290 | 296 | 261
U/L | 4 (60) | 2 (87) | 0 (63)

39. Secondary Outcome: Change From Baseline in Glucose
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 285 | 292 | 256
mmol/L | -0.09 (1.82) | 0.07 (1.95) | 0.17 (2.21)

40. Secondary Outcome: Change From Baseline in Urea
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 291 | 296 | 261
mmol/L | 0.1 (2.0) | 0.0 (2.3) | 0.0 (2.1)

41. Secondary Outcome: Change From Baseline in Blood Urea Nitrogen
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: milligrams per decilitre (mg/dL)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 291 | 296 | 261
milligrams per decilitre (mg/dL) | 0.1 (3.2) | 0.0 (3.7) | -0.1 (3.4)

42. Secondary Outcome: Change From Baseline in Creatinine
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: micromoles per litre (umol/L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 292 | 296 | 261
micromoles per litre (umol/L) | 2.7 (9.6) | 1.0 (11.1) | 1.7 (10.4)

43. Secondary Outcome: Change From Baseline in Bilirubin, Total
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 291 | 296 | 261
umol/L | 0.0 (4.5) | -0.1 (4.4) | 0.0 (4.0)

44. Secondary Outcome: Change From Baseline in Uric Acid
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 291 | 296 | 261
umol/L | 13.55 (78.13) | 1.03 (82.35) | 7.83 (88.05)

45. Secondary Outcome: Change From Baseline in Protein, Total
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: grams per litre (g/L)
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 291 | 296 | 261
grams per litre (g/L) | -1 (5) | -1 (5) | -1 (5)

46. Secondary Outcome: Change From Baseline in Albumin
Description: Week 48 - baseline
Time Frame: Baseline to Week 48 or at premature discontinuation if before Week 48
Population: Safety Set
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 291 | 296 | 261
g/L | 1 (4) | 1 (4) | 1 (4)

47. Secondary Outcome: Change From Baseline in Trough FEV1 After 2, 8, 16, 24, 32 and 40 Weeks
Description: Change From Baseline in Trough Forced Expiratory Volume in 1 second (FEV1) after 2, 8, 16, 24, 32 and 40 weeks. The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: as for outcome 1
Population: Full Analysis Set - Clinic Spirometry (FAS-PFT)
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 326 | 320 | 296
Litres
  Week 2 | 0.118 (0.011) | 0.133 (0.011) | 0.013 (0.012)
  Week 8 | 0.124 (0.012) | 0.150 (0.012) | -0.004 (0.013)
  Week 16 | 0.121 (0.013) | 0.125 (0.014) | -0.022 (0.014)
  Week 24 | 0.125 (0.013) | 0.121 (0.013) | -0.009 (0.013)
  Week 32 | 0.124 (0.013) | 0.132 (0.013) | -0.025 (0.014)
  Week 40 | 0.107 (0.013) | 0.133 (0.013) | -0.031 (0.014)

48. Secondary Outcome: Change From Baseline in Trough FVC After 2, 8, 16, 24, 32, 40 and 48 Weeks
Description: Change From Baseline in Trough Forced vital capacity (FVC) after 2, 8, 16, 24, 32, 40 and 48 weeks. The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: as for outcome 1
Population: Full Analysis Set - Clinic Spirometry (FAS-PFT)
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 326 | 320 | 296
Litres
  Week 2 | 0.163 (0.023) | 0.278 (0.024) | 0.025 (0.025)
  Week 8 | 0.168 (0.024) | 0.300 (0.024) | 0.009 (0.025)
  Week 16 | 0.145 (0.026) | 0.267 (0.027) | -0.019 (0.028)
  Week 24 | 0.155 (0.026) | 0.274 (0.026) | -0.012 (0.027)
  Week 32 | 0.156 (0.026) | 0.276 (0.026) | -0.038 (0.028)
  Week 40 | 0.130 (0.026) | 0.294 (0.027) | -0.043 (0.028)
  Week 48 | 0.108 (0.027) | 0.253 (0.027) | -0.070 (0.028)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry,centre and baseline value; Mean Difference (Final Values) = 0.178, Standard Error of Mean 0.039 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry,centre and baseline value; Mean Difference (Final Values) = 0.323, Standard Error of Mean 0.039 — Tiotropium Respimat 10mcg - Placebo

49. Secondary Outcome: Change From Baseline in FEV1 AUC0-3 After 2, 8, 16, 24, 32, 40 and 48 Weeks
Description: FEV1 AUC0-3 represents the Area under Curve over the time interval from 0 to 3 hours after 2, 8, 16, 24, 32, 40 and 48 weeks. The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: as for outcome 1
Population: Full Analysis Set - Clinic Spirometry (FAS-PFT)
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 326 | 320 | 296
Litres
  Week 2 | 0.256 (0.012) | 0.258 (0.012) | 0.045 (0.013)
  Week 8 | 0.246 (0.013) | 0.274 (0.013) | 0.041 (0.014)
  Week 16 | 0.241 (0.014) | 0.248 (0.014) | 0.024 (0.015)
  Week 24 | 0.242 (0.014) | 0.241 (0.014) | 0.026 (0.014)
  Week 32 | 0.239 (0.014) | 0.240 (0.014) | 0.019 (0.015)
  Week 40 | 0.225 (0.014) | 0.233 (0.014) | 0.003 (0.015)
  Week 48 | 0.212 (0.014) | 0.226 (0.014) | -0.008 (0.015)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry, centre and baseline value; Mean Difference (Final Values) = 0.220, Standard Error of Mean 0.021 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry, centre and baseline value; Mean Difference (Final Values) = 0.234, Standard Error of Mean 0.021 — Tiotropium Respimat 10mcg - Placebo

50. Secondary Outcome: Change From Baseline in FVC AUC0-3 After 2, 8, 16, 24, 32, 40 and 48 Weeks
Description: FVC AUC0-3 represents the Area under Curve over the time interval from 0 to 3 hours after 2, 8, 16, 24, 32, 40 and 48 weeks. The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: as for outcome 1
Population: Full Analysis Set - Clinic Spirometry (FAS-PFT)
Measure: Mean (Standard Error); unit: Litres
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 326 | 320 | 296
Litres
  Week 2 | 0.421 (0.024) | 0.492 (0.024) | 0.130 (0.025)
  Week 8 | 0.397 (0.026) | 0.538 (0.026) | 0.126 (0.027)
  Week 16 | 0.376 (0.028) | 0.487 (0.028) | 0.076 (0.029)
  Week 24 | 0.364 (0.027) | 0.465 (0.027) | 0.067 (0.029)
  Week 32 | 0.357 (0.028) | 0.465 (0.028) | 0.049 (0.029)
  Week 40 | 0.328 (0.028) | 0.453 (0.028) | 0.034 (0.029)
  Week 48 | 0.312 (0.028) | 0.422 (0.028) | 0.003 (0.029)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry, centre and baseline value; Mean Difference (Final Values) = 0.310, Standard Error of Mean 0.041 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, smoking status at entry, centre and baseline value; Mean Difference (Final Values) = 0.419, Standard Error of Mean 0.041 — Tiotropium Respimat 10mcg - Placebo

51. Secondary Outcome: Weekly Mean Morning Pre-dose PEFRs
Description: Weekly mean morning pre-dose peak expiratory flow rates (PEFRs). The means are adjusted for centre, smoking status at entry, and baseline value.
Time Frame: Weeks 2, 8, 16, 24, 32, 40, 48
Population: Full Analysis Set - Diary (FAS-DRY)
Measure: Mean (Standard Error); unit: Litres/minute
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 323 | 323 | 293
Litres/minute
  Week 2 | 255.4 (1.8) | 261.5 (1.8) | 235.4 (1.9)
  Week 8 | 259.0 (2.5) | 265.6 (2.5) | 241.8 (2.7)
  Week 16 | 262.7 (3.0) | 269.0 (3.0) | 241.1 (3.1)
  Week 24 | 265.7 (3.2) | 270.1 (3.2) | 244.3 (3.3)
  Week 32 | 267.2 (3.4) | 275.1 (3.4) | 244.7 (3.6)
  Week 40 | 267.0 (3.4) | 276.7 (3.4) | 247.4 (3.6)
  Week 48 | 268.5 (3.6) | 279.0 (3.6) | 245.9 (3.8)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = 22.5, Standard Error of Mean 5.3 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = 33.1, Standard Error of Mean 5.3 — Tiotropium Respimat 10mcg - Placebo

52. Secondary Outcome: Weekly Mean Evening PEFRs
Description: Weekly mean evening peak expiratory flow rates (PEFRs). The means are adjusted for centre, smoking status at entry, and baseline value.
Time Frame: Weeks 2, 8, 16, 24, 32, 40, 48
Population: Full Analysis Set - Diary (FAS-DRY)
Measure: Mean (Standard Error); unit: Litres/minute
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 323 | 322 | 293
Litres/minute
  Week 2 | 270.6 (2.0) | 279.2 (2.0) | 249.3 (2.1)
  Week 8 | 274.5 (2.7) | 282.1 (2.7) | 253.4 (2.9)
  Week 16 | 278.0 (3.1) | 284.1 (3.1) | 252.7 (3.2)
  Week 24 | 280.0 (3.3) | 287.0 (3.3) | 254.7 (3.4)
  Week 32 | 281.8 (3.4) | 290.6 (3.4) | 255.0 (3.6)
  Week 40 | 283.1 (3.6) | 292.2 (3.6) | 257.1 (3.7)
  Week 48 | 282.5 (3.9) | 292.5 (3.9) | 257.0 (4.1)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = 25.5, Standard Error of Mean 5.6 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = 35.5, Standard Error of Mean 5.6 — Tiotropium Respimat 10mcg - Placebo

53. Secondary Outcome: Weekly Mean Number of Puffs of Rescue Medication Per Day
Description: Weekly mean number of puffs of rescue medication used per day as required (PRN salbutamol). The means are adjusted for centre, smoking status at entry, and baseline value.
Time Frame: Weeks 2, 8, 16, 24, 32, 40, 48
Population: Full Analysis Set - Diary (FAS-DRY)
Measure: Mean (Standard Error); unit: Puffs
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 324 | 323 | 293
Puffs
  Week 2 | 1.9 (0.1) | 1.9 (0.1) | 2.7 (0.1)
  Week 8 | 2.0 (0.1) | 2.0 (0.1) | 2.7 (0.1)
  Week 16 | 2.1 (0.1) | 2.0 (0.1) | 2.8 (0.1)
  Week 24 | 2.1 (0.1) | 2.2 (0.1) | 3.0 (0.1)
  Week 32 | 2.2 (0.1) | 2.2 (0.1) | 3.0 (0.1)
  Week 40 | 2.2 (0.1) | 2.2 (0.1) | 3.0 (0.1)
  Week 48 | 2.3 (0.1) | 2.2 (0.1) | 3.1 (0.1)
Statistical Analysis 1: Comparison: Tiotropium Respimat 5mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = -0.8, Standard Error of Mean 0.2 — Tiotropium Respimat 5mcg - Placebo
Statistical Analysis 2: Comparison: Tiotropium Respimat 10mcg vs Placebo; Analysis for week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA analysis with terms for treatment, centre,smoking status at entry and baseline value; Mean Difference (Final Values) = -0.9, Standard Error of Mean 0.2 — Tiotropium Respimat 10mcg - Placebo

54. Secondary Outcome: Mahler TDI Scores
Description: Mahler Transitional Dyspnoea Index (TDI) scores measured as change in functional impairment, change in magnitude of tasks and change in magnitude of efforts over the treatment period. The means are adjusted for centre, smoking status at entry and baseline value.
  Worst score = -3, best score = +3
Time Frame: Week 48
Population: Full Analysis Set - Transitional Dyspnoea Index (FAS-TDI)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 318 | 313 | 273
Points on a scale
  Functional Impairment | 0.606 (0.049) | 0.679 (0.050) | 0.255 (0.053)
  Magnitude of Task | 0.650 (0.052) | 0.673 (0.052) | 0.291 (0.056)
  Magnitude of Effort | 0.633 (0.056) | 0.706 (0.056) | 0.240 (0.060)

55. Secondary Outcome: Saint George's Respiratory Questionnaire (SGRQ) Scores
Description: Saint George's Respiratory Questionnaire (SGRQ) Scores impacts, activities and symptoms. Worst score = 100, best score = 0.
  The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: Week 48
Population: Full Analysis Set - Saint George's Respiratory Questionnaire (FAS-QOL)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 318 | 315 | 275
Points on a scale
  Symptoms | 42.323 (1.064) | 41.798 (1.070) | 47.835 (1.146)
  Activities | 56.317 (0.823) | 55.180 (0.828) | 58.629 (0.887)
  Impacts | 29.413 (0.743) | 28.054 (0.747) | 32.466 (0.801)

56. Secondary Outcome: COPD Symptoms Scores
Description: COPD symptoms Scores - wheezing, shortness of breath, coughing and tightness of chest over the treatment period. Scale: 0 = None, 1 = Mild, 2 = Moderate, 3 = Severe
  The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: Week 48
Population: Full Analysis Set - COPD symptoms (FAS-SYM)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 326 | 321 | 295
Points on a scale
  Wheezing | 0.67 (0.04) | 0.65 (0.04) | 0.91 (0.04)
  Shortness of Breath | 1.35 (0.04) | 1.31 (0.04) | 1.51 (0.04)
  Coughing | 1.05 (0.04) | 1.04 (0.04) | 1.21 (0.04)
  Tightness of Chest | 0.61 (0.04) | 0.50 (0.04) | 0.78 (0.04)

57. Secondary Outcome: PGE Scores
Description: Physician's Global evaluation (PGE) scores over the treatment period. Scale: 1-2 = Poor, 3-4 = Fair, 5-6 = Good, 7-8 = Excellent
  The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: Week 48
Population: Full Analysis Set - Physician's Global Evaluation (FAS-PGE)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 327 | 322 | 295
Points on a scale | 5.18 (0.06) | 5.18 (0.06) | 4.62 (0.06)

58. Secondary Outcome: PGR Score
Description: Patient's Global rating (PGR) score over the treatment period. Scale: 1=much better to 7=much worse
  The means are adjusted for centre, smoking status at entry and baseline value.
Time Frame: Week 48
Population: Full Analysis Set - Patient's Global Rating (FAS-PGR)
Measure: Mean (Standard Error); unit: Points on a scale
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Number analyzed (Participants) | 319 | 316 | 276
Points on a scale | 3.05 (0.07) | 2.86 (0.07) | 3.52 (0.08)

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug administration.
Arm/Group | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Serious Adverse Events (participants affected / at risk) | 45 | 53 | 54
Other Adverse Events (participants affected / at risk) | 147 | 160 | 145
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Anaemia (Blood and lymphatic system disorders) | 0/332 | 1/332 | 0/319
Coagulopathy (Blood and lymphatic system disorders) | 0/332 | 1/332 | 0/319
Angina pectoris (Cardiac disorders) | 2/332 | 1/332 | 1/319
Angina unstable (Cardiac disorders) | 0/332 | 1/332 | 0/319
Atrial fibrillation (Cardiac disorders) | 1/332 | 1/332 | 1/319
Atrial flutter (Cardiac disorders) | 0/332 | 1/332 | 0/319
Cardiac failure (Cardiac disorders) | 3/332 | 0/332 | 0/319
Cardiac failure congestive (Cardiac disorders) | 1/332 | 1/332 | 1/319
Coronary artery disease (Cardiac disorders) | 1/332 | 0/332 | 1/319
Coronary artery insufficiency (Cardiac disorders) | 0/332 | 1/332 | 0/319
Myocardial infarction (Cardiac disorders) | 1/332 | 0/332 | 3/319
Pericardial effusion (Cardiac disorders) | 1/332 | 0/332 | 0/319
Ventricular tachycardia (Cardiac disorders) | 0/332 | 1/332 | 0/319
Cataract (Eye disorders) | 1/332 | 1/332 | 0/319
Retinal tear (Eye disorders) | 0/332 | 1/332 | 0/319
Abdominal pain (Gastrointestinal disorders) | 1/332 | 0/332 | 0/319
Colonic polyp (Gastrointestinal disorders) | 0/332 | 0/332 | 1/319
Gastritis (Gastrointestinal disorders) | 0/332 | 1/332 | 0/319
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/332 | 0/332 | 2/319
Haemorrhoids (Gastrointestinal disorders) | 0/332 | 1/332 | 0/319
Ileus (Gastrointestinal disorders) | 0/332 | 1/332 | 0/319
Inguinal hernia (Gastrointestinal disorders) | 0/332 | 3/332 | 0/319
Intestinal obstruction (Gastrointestinal disorders) | 0/332 | 0/332 | 1/319
Oesophageal haemorrhage (Gastrointestinal disorders) | 1/332 | 0/332 | 0/319
Rectocele (Gastrointestinal disorders) | 0/332 | 1/332 | 0/319
Adverse drug reaction (General disorders) | 0/332 | 1/332 | 0/319
Asthenia (General disorders) | 1/332 | 1/332 | 0/319
Chest pain (General disorders) | 1/332 | 0/332 | 1/319
Death (General disorders) | 0/332 | 5/332 | 2/319
Non-cardiac chest pain (General disorders) | 0/332 | 1/332 | 0/319
Pain (General disorders) | 0/332 | 0/332 | 1/319
Bile duct stone (Hepatobiliary disorders) | 0/332 | 0/332 | 1/319
Cholecystitis acute (Hepatobiliary disorders) | 0/332 | 1/332 | 0/319
Cholelithiasis (Hepatobiliary disorders) | 0/332 | 1/332 | 2/319
Drug hypersensitivity (Immune system disorders) | 0/332 | 0/332 | 1/319
Aspergillosis (Infections and infestations) | 0/332 | 0/332 | 1/319
Bronchial infection (Infections and infestations) | 0/332 | 0/332 | 1/319
Bronchitis (Infections and infestations) | 0/332 | 1/332 | 0/319
Bronchitis acute (Infections and infestations) | 0/332 | 0/332 | 1/319
Bronchopneumonia (Infections and infestations) | 1/332 | 0/332 | 0/319
Cellulitis (Infections and infestations) | 0/332 | 1/332 | 2/319
Diverticulitis (Infections and infestations) | 0/332 | 1/332 | 0/319
Gastroenteritis (Infections and infestations) | 1/332 | 0/332 | 1/319
Lobar pneumonia (Infections and infestations) | 0/332 | 0/332 | 2/319
Lower respiratory tract infection (Infections and infestations) | 1/332 | 0/332 | 0/319
Pneumonia (Infections and infestations) | 6/332 | 4/332 | 0/319
Respiratory tract infection (Infections and infestations) | 0/332 | 0/332 | 1/319
Sepsis (Infections and infestations) | 0/332 | 0/332 | 1/319
Superinfection lung (Infections and infestations) | 0/332 | 0/332 | 1/319
Urosepsis (Infections and infestations) | 0/332 | 0/332 | 1/319
Cardiac pacemaker malfunction (Injury, poisoning and procedural complications) | 1/332 | 0/332 | 0/319
Clavicle fracture (Injury, poisoning and procedural complications) | 0/332 | 0/332 | 1/319
Concussion (Injury, poisoning and procedural complications) | 1/332 | 0/332 | 0/319
Femur fracture (Injury, poisoning and procedural complications) | 1/332 | 0/332 | 1/319
Hip fracture (Injury, poisoning and procedural complications) | 0/332 | 0/332 | 1/319
Humerus fracture (Injury, poisoning and procedural complications) | 1/332 | 0/332 | 1/319
Joint dislocation (Injury, poisoning and procedural complications) | 0/332 | 0/332 | 1/319
Ligament injury (Injury, poisoning and procedural complications) | 0/332 | 1/332 | 0/319
Neck injury (Injury, poisoning and procedural complications) | 0/332 | 0/332 | 1/319
Tendon rupture (Injury, poisoning and procedural complications) | 0/332 | 1/332 | 0/319
Dehydration (Metabolism and nutrition disorders) | 0/332 | 1/332 | 0/319
Hypoglycaemia (Metabolism and nutrition disorders) | 0/332 | 0/332 | 1/319
Back pain (Musculoskeletal and connective tissue disorders) | 0/332 | 1/332 | 0/319
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0/332 | 0/332 | 1/319
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0/332 | 1/332 | 0/319
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2/332 | 0/332 | 0/319
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/332 | 1/332 | 0/319
Bladder cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/332 | 1/332 | 0/319
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/332 | 0/332 | 0/319
Bronchioloalveolar carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/332 | 0/332 | 0/319
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/332 | 1/332 | 0/319
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/332 | 0/332 | 1/319
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/332 | 0/332 | 1/319
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/332 | 0/332 | 1/319
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/332 | 0/332 | 0/319
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/332 | 0/332 | 0/319
Oesophageal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/332 | 1/332 | 0/319
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/332 | 1/332 | 2/319
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/332 | 0/332 | 0/319
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/332 | 0/332 | 1/319
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/332 | 0/332 | 0/319
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/332 | 1/332 | 0/319
Cerebral infarction (Nervous system disorders) | 0/332 | 1/332 | 0/319
Cerebrovascular accident (Nervous system disorders) | 0/332 | 1/332 | 2/319
Dysarthria (Nervous system disorders) | 1/332 | 0/332 | 0/319
Facial paresis (Nervous system disorders) | 0/332 | 0/332 | 1/319
Guillain-Barre syndrome (Nervous system disorders) | 0/332 | 1/332 | 0/319
Ischaemic stroke (Nervous system disorders) | 0/332 | 1/332 | 0/319
Normal pressure hydrocephalus (Nervous system disorders) | 1/332 | 0/332 | 0/319
Sciatica (Nervous system disorders) | 1/332 | 0/332 | 0/319
Syncope (Nervous system disorders) | 0/332 | 0/332 | 1/319
Aggression (Psychiatric disorders) | 0/332 | 0/332 | 1/319
Confusional state (Psychiatric disorders) | 2/332 | 0/332 | 0/319
Cystocele (Renal and urinary disorders) | 0/332 | 1/332 | 0/319
Haematuria (Renal and urinary disorders) | 0/332 | 1/332 | 0/319
Renal cyst (Renal and urinary disorders) | 0/332 | 1/332 | 0/319
Renal failure acute (Renal and urinary disorders) | 0/332 | 1/332 | 0/319
Urinary retention (Renal and urinary disorders) | 0/332 | 2/332 | 0/319
Urinary tract obstruction (Renal and urinary disorders) | 0/332 | 1/332 | 0/319
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0/332 | 1/332 | 0/319
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/332 | 0/332 | 0/319
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/332 | 1/332 | 0/319
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 13/332 | 11/332 | 17/319
Cough (Respiratory, thoracic and mediastinal disorders) | 0/332 | 1/332 | 0/319
Diaphragmatic hernia (Respiratory, thoracic and mediastinal disorders) | 0/332 | 1/332 | 0/319
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2/332 | 0/332 | 0/319
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1/332 | 1/332 | 1/319
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0/332 | 0/332 | 1/319
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0/332 | 0/332 | 1/319
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1/332 | 0/332 | 0/319
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1/332 | 0/332 | 1/319
Eczema (Skin and subcutaneous tissue disorders) | 1/332 | 0/332 | 0/319
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0/332 | 0/332 | 1/319
Psoriasis (Skin and subcutaneous tissue disorders) | 1/332 | 0/332 | 0/319
Skin ulcer (Skin and subcutaneous tissue disorders) | 1/332 | 0/332 | 0/319
Deep vein thrombosis (Vascular disorders) | 0/332 | 1/332 | 0/319
Hypertension (Vascular disorders) | 0/332 | 1/332 | 0/319
Hypotension (Vascular disorders) | 0/332 | 0/332 | 1/319
Peripheral vascular disorder (Vascular disorders) | 0/332 | 1/332 | 0/319
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Tiotropium Respimat 5mcg | Tiotropium Respimat 10mcg | Placebo
Dry mouth (Gastrointestinal disorders) | 15/332 | 44/332 | 4/319
Nasopharyngitis (Infections and infestations) | 41/332 | 31/332 | 30/319
Back pain (Musculoskeletal and connective tissue disorders) | 18/332 | 13/332 | 15/319
Chronic obstructive airways disease exacerbated (Respiratory, thoracic and mediastinal disorders) | 95/332 | 94/332 | 114/319
Cough (Respiratory, thoracic and mediastinal disorders) | 14/332 | 16/332 | 16/319

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.